CLINICAL TRIAL: NCT04288232
Title: A Multicenter, Open-label, Prospective, Interventional Study to Assess the Efficacy and Safety of Aflibercept as Mono-therapy in Treat and Extend Regimen for DME Patients in Taiwan
Brief Title: Efficacy and Safety of Aflibercept as Mono-therapy in Treat and Extend Regimen for DME Patients in Taiwan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Kaohsiung Veterans General Hospital. (Other); National Taiwan University Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17683
Record Dates: First submitted 2020-02-09; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Center-involved Diabetic Macular Edema
Keywords: anti-VEGF; intravitreal aflibercept; diabetic macular edema; Treat-and-Extend regimen
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravitreal aflibercept (Experimental): Intravitreal injection of aflibercept 2.0mg/0.05 ml Aflibercept was administered with 5 monthly loadings followed by treat-and-extend with a 4-week interval increment/decrement with maxima cap at 12 weeks to visual/anatomic stability.
  Interventions: Drug: Aflibercept Injection [Eylea]

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — Intravitreal aflibercept Injection 2.0mg/0.05 ml

SUMMARY:
Phase IIIb, multicenter, open-label, prospective, interventional study to assess the potential benefit of Aflibercept treatment administered IVT at a dosage of 2 mg with five monthly loading doses and then treat and extend over 48 weeks, with the primary endpoint as BCVA assessed at Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 20 years old with type 1 or 2 diabetes mellitus
* Subjects with DME secondary to diabetes mellitus involving the center of the macula (defined as the area of the center subfield of optical coherence tomography [OCT]) in the study eye
* Retinal thickness as assessed by OCT above (>) 300 um in the study eye
* BCVA ETDRS letter score of 73 to 24 (20/40 to 20/320) in the study eye
* Would be able to comply with clinic visits and study-related procedures
* Would be able to provide a signed informed consent form (ICF)

Exclusion Criteria:

1. Ocular conditions with a poorer prognosis in the fellow eye than in the study eye
2. History of vitreoretinal surgery and/or including scleral buckling in the study eye
3. Laser photocoagulation (pan-retinal or macular) in the study eye within 90 days of Day 1
4. Against the background of a relevant number of previous macular laser treatments the investigator's point of view was that the subjects had no potential to benefit from laser treatments (e.g., if too many laser treatments were applied in the past)
5. Previous use of intraocular or periocular corticosteroids in the study eye within 120 days of Day 1
6. Previous treatment with anti-angiogenic drugs in either eye (pegaptanib sodium, bevacizumab, ranibizumab etc.) within 90 days of Day 1
7. High risk proliferative diabetic retinopathy (PDR) in the study eye upon physician's discretion

   High risk = the presence of any of the following:
   * Vitreous hemorrhage
   * New vessels on the disk >1/3 disk diameter
   * New vessels elsewhere >1/2 disk diameter
8. History of idiopathic or autoimmune uveitis in the study eye
9. Cataract surgery within 90 days before Day 1 in the study eye
10. Aphakia in the study eye
11. Yttrium-aluminium-garnet (YAG) capsulotomy in the study eye within 30 days before Day 1
12. Any other intraocular surgery within 90 days of Day 1 in the study eye
13. Vitreomacular traction or epiretinal membrane in the study eye evident biomicroscopically or on OCT that is thought to affect central vision
14. Current iris neovascularization, vitreous hemorrhage, or tractional retinal detachment in the study eye
15. Pre-retinal fibrosis involving the macula in the study eye
16. Structural damage to the center of the macula in the study eye that was likely to preclude improvement in BCVA following the resolution of macular edema including atrophy of the retinal pigment epithelium, subretinal fibrosis or scar, significant macular ischemia or organized hard exudates
17. Ocular inflammation including trace or above in the study eye
18. Evidence of infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye
19. Filtration surgery for glaucoma in the past or likely to be needed in the future on the study eye
20. Intraocular pressure (IOP) ≥ 25 mmHg in the study eye
21. High myopia (≤ -6.0 diopters or axial length of ≥26.5 mm) prior to any possible refractive or cataract surgery
22. Concurrent disease in the study eye, other than DME, that could compromise VA, require medical or surgical intervention during the study period, or could confound interpretation of the results (including retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization of any cause)
23. Only 1 functional eye even if that eye was otherwise eligible for the study
24. Ocular media of insufficient quality to obtain fundus and OCT images
25. Current treatment for a serious systemic infection
26. Administration of systemic anti-angiogenic agents within 180 days before Day 1
27. Uncontrolled diabetes mellitus, as defined by Hemoglobin A1c; (glycosylated hemoglobin) (HbA1c)>10%.
28. Uncontrolled blood pressure (defined as systolic >160 mmHg or diastolic >95 mmHg while subject was sitting)
29. History of either cerebral vascular accident and/or myocardial infarction within 180 days prior to Day 1
30. Renal failure requiring dialysis or renal transplant
31. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, might affect interpretation of the results of the study, or rendered the subject at high risk for treatment complications
32. Pregnant or breast-feeding women
33. Sexually active men or women of childbearing potential who were unwilling to practice adequate contraception during the study were excluded (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly or diaphragm plus contraceptive sponge, foam, or jelly).
34. Allergy to fluorescein
35. Participation in an investigational study within 30 days prior to screening visit that involved treatment with any drug (excluding vitamins and minerals) or device

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Mean change of best corrected visual acuity (BCVA) from baseline to week 52 | baseline to week 52
  BCVA is measured by ETDRS chart

SECONDARY OUTCOMES:
Mean change in central subfoveal thickness (CST) from baseline to week 52. | baseline to week 52
  Central subfoveal thickness (CST) as assessed by OCT
Mean/medium number of injection from baseline to week 52 | baseline to week 52
  Mean/medium number of intravitreal aflibercept injection from baseline to week 52
Proportion of subjects who gained > 15 ETDRS letters from baseline to week 52 | baseline to week 52
  BCVA is measured by ETDRS chart
Proportion of subjects with > 2-step improvement in DRSS from baseline to week 52 | baseline to week 52
  DR level as assessed by diabetic retinopathy severity score (DRSS)
Proportion of subjects demonstrating retina dry at week 20 and week 52 | week 20 and week 52
  Retina dry as assessed by OCT

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Jen Chen, MD, PhD, Principal Investigator — Department of Ophthalmology, Taipei Veterans General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. III. Prevalence and risk of diabetic retinopathy when age at diagnosis is 30 or more years. Arch Ophthalmol. 1984 Apr;102(4):527-32. doi: 10.1001/archopht.1984.01040030405011. PMID 6367725
- [Background] Moss SE, Klein R, Klein BE. Ten-year incidence of visual loss in a diabetic population. Ophthalmology. 1994 Jun;101(6):1061-70. doi: 10.1016/s0161-6420(94)31217-6. PMID 8008348
- [Background] Moss SE, Klein R, Klein BE. The 14-year incidence of visual loss in a diabetic population. Ophthalmology. 1998 Jun;105(6):998-1003. doi: 10.1016/S0161-6420(98)96025-0. PMID 9627648
- [Background] Zhang X, Saaddine JB, Chou CF, Cotch MF, Cheng YJ, Geiss LS, Gregg EW, Albright AL, Klein BE, Klein R. Prevalence of diabetic retinopathy in the United States, 2005-2008. JAMA. 2010 Aug 11;304(6):649-56. doi: 10.1001/jama.2010.1111. PMID 20699456
- [Background] Yang W, Lu J, Weng J, Jia W, Ji L, Xiao J, Shan Z, Liu J, Tian H, Ji Q, Zhu D, Ge J, Lin L, Chen L, Guo X, Zhao Z, Li Q, Zhou Z, Shan G, He J; China National Diabetes and Metabolic Disorders Study Group. Prevalence of diabetes among men and women in China. N Engl J Med. 2010 Mar 25;362(12):1090-101. doi: 10.1056/NEJMoa0908292. PMID 20335585
- [Background] Wang FH, Liang YB, Zhang F, Wang JJ, Wei WB, Tao QS, Sun LP, Friedman DS, Wang NL, Wong TY. Prevalence of diabetic retinopathy in rural China: the Handan Eye Study. Ophthalmology. 2009 Mar;116(3):461-7. doi: 10.1016/j.ophtha.2008.10.003. Epub 2009 Jan 24. PMID 19168222
- [Background] Ferrara N, Davis-Smyth T. The biology of vascular endothelial growth factor. Endocr Rev. 1997 Feb;18(1):4-25. doi: 10.1210/edrv.18.1.0287. No abstract available. PMID 9034784
- [Background] Ferrara N. VEGF: an update on biological and therapeutic aspects. Curr Opin Biotechnol. 2000 Dec;11(6):617-24. doi: 10.1016/s0958-1669(00)00153-1. PMID 11102799
- [Background] Nguyen QD, Tatlipinar S, Shah SM, Haller JA, Quinlan E, Sung J, Zimmer-Galler I, Do DV, Campochiaro PA. Vascular endothelial growth factor is a critical stimulus for diabetic macular edema. Am J Ophthalmol. 2006 Dec;142(6):961-9. doi: 10.1016/j.ajo.2006.06.068. Epub 2006 Aug 2. PMID 17046701
- [Background] Bhagat N, Grigorian RA, Tutela A, Zarbin MA. Diabetic macular edema: pathogenesis and treatment. Surv Ophthalmol. 2009 Jan-Feb;54(1):1-32. doi: 10.1016/j.survophthal.2008.10.001. PMID 19171208
- [Background] Grover D, Li TJ, Chong CC. Intravitreal steroids for macular edema in diabetes. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD005656. doi: 10.1002/14651858.CD005656.pub2. PMID 18254088
- [Background] El Sanharawi M, Kowalczuk L, Touchard E, Omri S, de Kozak Y, Behar-Cohen F. Protein delivery for retinal diseases: from basic considerations to clinical applications. Prog Retin Eye Res. 2010 Nov;29(6):443-65. doi: 10.1016/j.preteyeres.2010.04.001. Epub 2010 Apr 14. PMID 20398784
- [Background] Angelousi A, Larger E. Anaemia, a common but often unrecognized risk in diabetic patients: a review. Diabetes Metab. 2015 Feb;41(1):18-27. doi: 10.1016/j.diabet.2014.06.001. Epub 2014 Jul 17. PMID 25043174
- [Background] Buyukkaya E, Karakas MF, Karakas E, Akcay AB, Tanboga IH, Kurt M, Sen N. Correlation of neutrophil to lymphocyte ratio with the presence and severity of metabolic syndrome. Clin Appl Thromb Hemost. 2014 Mar;20(2):159-63. doi: 10.1177/1076029612459675. Epub 2012 Sep 18. PMID 22992349
- [Background] Sefil F, Ulutas KT, Dokuyucu R, Sumbul AT, Yengil E, Yagiz AE, Yula E, Ustun I, Gokce C. Investigation of neutrophil lymphocyte ratio and blood glucose regulation in patients with type 2 diabetes mellitus. J Int Med Res. 2014 Apr;42(2):581-8. doi: 10.1177/0300060513516944. Epub 2014 Feb 24. PMID 24567354
- [Result] Arevalo JF, Sanchez JG, Wu L, Maia M, Alezzandrini AA, Brito M, Bonafonte S, Lujan S, Diaz-Llopis M, Restrepo N, Rodriguez FJ, Udaondo-Mirete P; Pan-American Collaborative Retina Study Group. Primary intravitreal bevacizumab for diffuse diabetic macular edema: the Pan-American Collaborative Retina Study Group at 24 months. Ophthalmology. 2009 Aug;116(8):1488-97, 1497.e1. doi: 10.1016/j.ophtha.2009.03.016. Epub 2009 Jul 9. PMID 19545900
- [Result] Diabetic Retinopathy Clinical Research Network; Elman MJ, Aiello LP, Beck RW, Bressler NM, Bressler SB, Edwards AR, Ferris FL 3rd, Friedman SM, Glassman AR, Miller KM, Scott IU, Stockdale CR, Sun JK. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2010 Jun;117(6):1064-1077.e35. doi: 10.1016/j.ophtha.2010.02.031. Epub 2010 Apr 28. PMID 20427088
- [Result] Do DV, Nguyen QD, Boyer D, Schmidt-Erfurth U, Brown DM, Vitti R, Berliner AJ, Gao B, Zeitz O, Ruckert R, Schmelter T, Sandbrink R, Heier JS; da Vinci Study Group. One-year outcomes of the da Vinci Study of VEGF Trap-Eye in eyes with diabetic macular edema. Ophthalmology. 2012 Aug;119(8):1658-65. doi: 10.1016/j.ophtha.2012.02.010. Epub 2012 Apr 24. PMID 22537617
- [Result] Korobelnik JF, Do DV, Schmidt-Erfurth U, Boyer DS, Holz FG, Heier JS, Midena E, Kaiser PK, Terasaki H, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Brown DM. Intravitreal aflibercept for diabetic macular edema. Ophthalmology. 2014 Nov;121(11):2247-54. doi: 10.1016/j.ophtha.2014.05.006. Epub 2014 Jul 8. PMID 25012934
- [Result] Terasaki H, Shiraki K, Ohji M, Metzig C, Schmelter T, Zeitz O, Sowade O, Kobayashi M, Vitti R, Berliner A, Shiraga F. EFFICACY AND SAFETY OUTCOMES OF INTRAVITREAL AFLIBERCEPT FOCUSING ON PATIENTS WITH DIABETIC MACULAR EDEMA FROM JAPAN. Retina. 2019 May;39(5):938-947. doi: 10.1097/IAE.0000000000002100. PMID 29470308
- [Derived] Sheu SJ, Yang CH, Lai CC, Wu PC, Chen SJ. One-year outcomes of the treat-and-extend regimen using aflibercept for the treatment of diabetic macular edema. J Chin Med Assoc. 2022 Feb 1;85(2):246-251. doi: 10.1097/JCMA.0000000000000680. PMID 34974510